CLINICAL TRIAL: NCT05800509
Title: Gestational Diabetes and Depression in Pregnancy and the Postpartum Period Among Primipara Women: A Longitudinal Study and Interventive Program
Brief Title: Gestational Diabetes and Perinatal Depression: an Intervention Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Mackay Memorial Hospital (Other); Taiwan Adventist Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202103014RINC
Record Dates: First submitted 2023-02-07; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-02

CONDITIONS: Gestational Diabetes Mellitus; Postpartum Depression; Perinatal Depression
Keywords: Antepartum Depression; Gestational Diabetes Mellitus; Perinatal Depression; Postpartum Depression; Health Interventions
MeSH Terms: conditions — Diabetes, Gestational; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: This study is randomized-controlled trial, half of enrolled participants acquire the intervention of health education and regular health service from hospital, another half only acquire regular health service from hospital.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The participants and their partners will receive structured questionnaires respectively at 22nd and 35th week of pregnancy, and 3rd month and 6th month after delivery. The context of questionnaire includes basic information (age, level of education and occupation of the participant and her partner, household income, and status of marriage), marriage satisfaction, obstetrics and gynecological history (history of abortion, intended pregnancy , and artificial insemination), psychiatric history, family history of diabetes mellitus, height, pre-pregnancy weight, sleeping status, and basic knowledge of gestational diabetes mellitus.
  A website of health education of gestational diabetes mellitus with several short clips of health education (maternity management/counseling, healthy lifestyles, partner support...etc) for participants and their partners will be given right after the questionnaire of 22nd week of pregnancy received from the participants and their partners.
  Interventions: Behavioral: Clips Intervention
- Controlled group (Sham Comparator): The participants and their partners will receive structured questionnaires respectively at 22nd and 35th week of pregnancy, and 3rd month and 6th month after delivery. The context of questionnaire includes basic information (age, level of education and occupation of the participant and her partner, household income, and status of marriage), marriage satisfaction, obstetrics and gynecological history (history of abortion, intended pregnancy , and artificial insemination), psychiatric history, family history of diabetes mellitus, height, pre-pregnancy weight, sleeping status, and basic knowledge of gestational diabetes mellitus.
  A website of health education about gestational diabetes mellitus for participants and their partners will be given right after the questionnaire of 22nd week of pregnancy received from the participants and their partners.
  Interventions: Device: Structured Questionnaire Only

INTERVENTIONS:
Behavioral: Clips Intervention — A website of health education of gestational diabetes mellitus with several short clips of health education (maternity management/counseling, healthy lifestyles, partner support...etc) for participants and their partners will be given right after the questionnaire of 22nd week of pregnancy received from the participants and their partners. There are pretest and posttest questions on the structured questionnaires of 22nd week and 35th week of pregnancy and 3rd month after delivery.
  Arms: Experimental Group
Device: Structured Questionnaire Only — A website of health education about gestational diabetes mellitus will be given to participants and their partners, then structured questionnaires and regular health service from the hospital continue to be given.
  Arms: Controlled group

SUMMARY:
Background: The gestational diabetes mellitus and perinatal depression are both global public health issues with high prevalence. Non-perinatal diabetes mellitus and depression are confirmed to have reciprocal influence, which is bidirectional relationship. However, there are still no any confirmations of relationship in the perinatal period. The reason could be that these kinds of studies mostly had been done for postpartum depression, they had rarely been discussed with a clearly sequential influence between gestational diabetes mellitus and perinatal depression. Additionally, there have not been so many Asian countries which been done this kind of studies, therefore, this study will focus on the relationship of primiparous gestational diabetes mellitus and perinatal depression.

Purpose: This study will discuss the bidirectional relationship of gestational diabetes mellitus and perinatal depression. In the other words, the prenatal depression influences on gestational diabetes mellitus, and vice versa. Those changeable factors, such as social support, health behavior, prenatal body index, weight gain during pregnancy, perinatal complications…etc, will be tested for whether they could be regulators or not between the gestational diabetes mellitus and perinatal depression.Afterwards, a part of participants with diagnosis of gestational diabetes mellitus will receive the intervention of health education to influence the health behavior, then depression and other obstetrics and gynecological results will be tested for effects.

DETAILED DESCRIPTION:
Background: The gestational diabetes mellitus and perinatal depression are both global public health issues with high prevalence. Non-perinatal diabetes mellitus and depression are confirmed to have reciprocal influence, which is bidirectional relationship. However, there are still no any confirmations of relationship in the perinatal period. The reason could be that these kinds of studies mostly had been done for postpartum depression, they had rarely been discussed with a clearly sequential influence between gestational diabetes mellitus and perinatal depression. Additionally, there have not been so many Asian countries which been done this kind of studies, therefore, this study will focus on the relationship of primiparous gestational diabetes mellitus and perinatal depression.

Purpose: This study will discuss the bidirectional relationship of gestational diabetes mellitus and perinatal depression. In the other words, the prenatal depression influences on gestational diabetes mellitus, and vice versa. Those changeable factors, such as social support, health behavior, prenatal body index, weight gain during pregnancy, perinatal complications…etc, will be tested for whether they could be regulators or not between the gestational diabetes mellitus and perinatal depression. Afterwards, a part of participants with diagnosis of gestational diabetes mellitus will receive the intervention of health education to influence the health behavior, then depression and other obstetrics and gynecological results will be tested for effects.

Method: The researchers will explain the purpose, procedure, and informed-consent of this study, then informed-consent form will be signed, and the structured questionnaire at 22nd week of pregnancy (including basic information (age, level of education and occupation of the participant and her partner, household income, and status of marriage), marriage satisfaction, obstetrics and gynecological history (history of abortion, intended pregnancy , and artificial insemination), psychiatric history, family history of diabetes mellitus, height, pre-pregnancy weight, sleeping status, and basic knowledge of gestational diabetes mellitus) will be given to fill out. The participants will be needed to record the value and date and time of blood sugar, and the picture of meals and snacks. After the first questionnaire is received from participants and their partners, a website of health education of gestational diabetes mellitus with several short clips of health education (maternity management/counseling, healthy lifestyles, partner support...etc) for participants and their partners of experimental group will be given. However, the participants and their partner of controlled group only receive a website of health education of gestational diabetes mellitus without any clips of health education. Afterward, structured questionnaire will be also given to the participants and their partners at 35th week of pregnancy, 3rd month and 6th months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* 1. The diagnosis of gestational diabetes mellitus.
* 2. The primiparous women.
* 3. No any history of disease* before the pregnancy or do have history of disease* without taking any medicines. (*disease, eg. hypertension, diabetes mellitus, hyperthyroidism...etc.)
* 4. No recurrent pregnancy loss and stable condition in the first trimester of pregnancy.
* 5. Using smart phone.
* 6. Being willing to participate in this study.

Exclusion Criteria:

- 1. No diagnosis of diabetes mellitus before pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women will be recruited at the hospitals, and then their partners (the role of partners as biological fathers during pregnancy) will be invited to participate this study.
Enrollment: 226 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants with interventional health education as accessed by the questionnaire of EPDS change from baseline within the period from 22nd week of pregnancy to 6 months after delivery. | From 22nd week of pregnancy to 6 months after delivery.
  Perinatal depression is measured by Edinburgh Postnatal Depression Scale (EPDS) in questionnaire.
Number and percentage of participants with interventional health education as accessed by the self-drafted questionnaire of social support change from baseline within the period from 22nd week of pregnancy to 6 months after delivery. | From 22nd week of pregnancy to 6 months after delivery.
  The social support scale is measured by self-drafted questionnaire, those questions are ranked within 5 intervals, from very insufficient to very sufficient.
Number and percentage of participants with interventional health education as accessed by the questionnaire of PPAQ change from baseline within the period from 22nd week of pregnancy to 6 months after delivery. | From 22nd week of pregnancy to 6 months after delivery.
  Physical activity is measured by Pregnancy Physical Activity Questionnaire (PPAQ) in questionnaire.
Number and percentage of participants with interventional health education as accessed by the self-drafted questionnaire of habit of diet change from baseline within the period from 22nd week of pregnancy to 6 months after delivery. | From 22nd week of pregnancy to 6 months after delivery.
  The habit of diet is measured by self-drafted questionnaire, those questions are related to frequencies of diet, preferences of diet, choices of diet.
Number and percentage of participants with interventional health education as accessed by the medical record of maternal body weight in kilograms change from baseline of pre-pregnancy within the 6 months after delivery. | From 22nd week of pregnancy to 6 months after delivery.
  The maternal body weight in kilograms is acquired from medical record.
Number and percentage of participants with interventional health education as accessed by the medical record of maternal BMI in kg/m^2 change from baseline of pre-pregnancy within the 6 months after delivery. | From 22nd week of pregnancy to 6 months after delivery.
  The maternal Body Mass Index (BMI) in kg/m^2 is calculated by body weight in kilograms and height in meters, which are acquired from medical record.
Number and percentage of participants with interventional health education as accessed by the questionnaire of knowledge and self-management of gestational diabetes mellitus change from baseline from 22nd week of pregnancy to 6 months after delivery. | From 22nd week of pregnancy to 6 months after delivery.
  The knowledge and self-management of gestational diabetes mellitus are measured by self-drafted questionnaire, which are true/false questions.
Number and percentage of participants with interventional health education as accessed by the self-drafted questionnaire of health belief change from baseline within the period from 22nd week of pregnancy to 6 months after delivery. | From 22nd week of pregnancy to 6 months after delivery.
  The health belief is measured by self-drafted questionnaire, those questions are ranked within 5 intervals, from extremely disagree to extremely agree.
Number and percentage of participants with interventional health education as accessed by the medical record of their perinatal complications. | From 22nd week of pregnancy to 6 months after delivery.
  The perinatal complication is acquired from medical record
Number and percentage of participants with interventional health education as accessed by the medical record of their infants' body weight in kilograms. | Within 6 months after delivery
  The infants' body weight in kilograms is acquired from medical record.

IPD SHARING:
Plan to Share IPD: No